CLINICAL TRIAL: NCT07201766
Title: The Efficacy of Intralesional Bleomycin as Compared to 5-Flourouracil (5-FU) and Triamcinolone Acetonide (TAC) for the Treatment of Keloids: A Randomized Control Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Shumaila Dogar, Consultant, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 645/RC/KEMU
Record Dates: First submitted 2025-09-19; First posted 2025-10-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Keloids Scars
Keywords: intralesional injection; bleomycin; keloid scars
MeSH Terms: conditions — Keloid | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Study Design: Randomized Control Trial Place of Study: Plastic Surgery department, Mayo Hospital Lahore Duration of Study: 6 months after approval of synopsis Sample Size: sample size of 104 patients (52 in each group) Sampling Technique Non probability consecutive sampling All, patients aged 13-60 years of age, either gender enrolled for Keloid treatment under local anaesthesia.
  Exclusion Criteria:
  Allergic to bleomycin, 5-FU DIABETICS VASCULAR INSUFFICIENCY AT THE AFFECTED SITE
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Efficacy of Intralesional Bleomycinin treatment of keloids (Experimental): Group B will be given injection Bleomycin 1.5 IU /ml (15 units vial dilution in 10ml Normal saline) 1 ml of this 1cm apart intralesionally as 0.1- 0.2ml/cm2 with max dose of 5ml per session and repeat after 2 weeks. Treatment will be given in two groups by a researcher blinded of the treatment being given in each group. POSAS patient and observer scar scale will be used to assess the keloids at 0, 2, 4, 6, 8, 10, and 12 weeks and during follow ups afterwards, assessments will be carried out by another researcher who will assess the improvement on the scale of 0-no improvement, to excellent-75-100% improvement in terms of POSAS variables.
  Interventions: Drug: intralesional bleomycin
- The Efficacy of 5-fluorouracil (5-FU) and Triamcinolone Acetonide in treatment of keloids (Experimental): Group A will be given 1ml if 0.9ml/22.5mg (25mg/ml) of 5-FU with 0.1 ml/4mg (40mg/ml) of Triamcinolone Acetonide, intralesionally 1cm apart, as 0.1- 0.2ml/cm2 with max dose of 5ml per session and repeat after every 2 weeks.
  Interventions: Drug: 5-flourouracil and triamcinolone acetonide

INTERVENTIONS:
Drug: intralesional bleomycin — The role of intralesional bleomycin for the treatment of keloids needs further establishment in terms of effective concentration, number of sessions and post treatment ulceration or/and hypopigmentation. Additionally, its comparison to the commonly used and proven, more effective combination than intralesional steroid alone i-e 5-FU in combination with the intralesional steroid, need also be done so that if found affective will be able to deal with the pathological scar as a 1 st line therapeutic drug. With a strong study design and an adequate sample size, and particularly in a specialized tertiary care clinical setup, Our study, seeks to get over the aforementioned limitations, and will delineates the appropriate guidelines for the management of these pathological scars, and suggest option with the best outcomes, as well as lesser side effects and recurrence rates.
  Arms: The Efficacy of Intralesional Bleomycinin treatment of keloids
Drug: 5-flourouracil and triamcinolone acetonide — The role of intralesional bleomycin for the treatment of keloids needs further establishment in terms of effective concentration, number of sessions and post treatment ulceration or/and hypopigmentation. Additionally, its comparison to the commonly used and proven, more effective combination than intralesional steroid alone i-e 5-FU in combination with the intralesional steroid, need also be done so that if found affective will be able to deal with the pathological scar as a 1 st line therapeutic drug. With a strong study design and an adequate sample size, and particularly in a specialized tertiary care clinical setup, Our study, seeks to get over the aforementioned limitations, and will delineates the appropriate guidelines for the management of these pathological scars, and suggest option with the best outcomes, as well as lesser side effects and recurrence rates.
  Arms: The Efficacy of 5-fluorouracil (5-FU) and Triamcinolone Acetonide in treatment of keloids

SUMMARY:
The goal of this clinical trial is to learn if drug bleomycin intralesionally is beneficial than intralesional 5FU and Triamcinolone Acetonide in treating Keloids. The main questions it aims to answer are:

Does drug Bleomycin injected intrasleisonally lower the time duration to effectively treat the keloids in participants as compared to intralesional Triamcinolone Acetonide and 5-Flourouracil? Researchers will compare drug Bleomycin and 5FU plus Triamcinolone Acetonide and determine if bleomycin is better.

Participants will:

Treatment will be given in two groups by a researcher blinded of the treatment being given in each group. POSAS patient and observer scar scale will be used to assess the keloids at 0, 2, 4, 6, 8, 10, and 12 weeks and during follow ups afterwards, assessments will be carried out by another researcher who will assess the improvement on the scale of 0-no improvement, to excellent-75-100% improvement in terms of POSAS variables. Effectiveness will be indicated by 50% reduction in POSAS score from the baseline.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if drug bleomycin intralesionally is beneficial than intralesional 5FU and Triamcinolone Acetonide in treating Keloids. The main questions it aims to answer are:

Does drug Bleomycin injected intrasleisonally lower the time duration to effectively treat the keloids in participants as compared to intralesional Triamcinolone Acetonide and 5-Flourouracil? Researchers will compare drug Bleomycin and 5FU plus Triamcinolone Acetonide and determine if bleomycin is better.

An informed, written consent will be taken from the patients. Clinical data including demographic data will be recorded. Patients will be randomly divided into two groups by using random allocation software 2.0. Group A will be given 1ml if 0.9ml/22.5mg (25mg/ml) of 5-FU with 0.1 ml/4mg (40mg/ml) of Triamcinolone Acetonide, intralesionally 1cm apart, as 0.1- 0.2ml/cm2 with max dose of 5ml per session and repeat after every 2 weeks. Group B will be given injection Bleomycin 1.5 IU /ml (15 units vial dilution in 10ml Normal saline) 1 ml of this 1cm apart intralesionally as 0.1- 0.2ml/cm2 with max dose of 5ml per session and repeat after 2 weeks. Treatment will be given in two groups by a researcher blinded of the treatment being given in each group. POSAS patient and observer scar scale will be used to assess the keloids at 0, 2, 4, 6, 8, 10, and 12 weeks and during follow ups afterwards, assessments will be carried out by another researcher who will assess the improvement on the scale of 0-no improvement, to excellent-75-100% improvement in terms of POSAS variables. Effectiveness will be indicated by 50% reduction in POSAS score from the baseline. All the data will be noted on a specially designed pro forma.

ELIGIBILITY:
Inclusion Criteria:

* All, patients aged 13-60 years of age, either gender enrolled for Keloid treatment under local anaesthesia.

Exclusion Criteria:

* Allergic to bleomycin, 5-FU DIABETICS VASCULAR INSUFFICIENCY AT THE AFFECTED SITE

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The Efficacy in terms of POSAS SCAR SCALE of Intralesional Bleomycin as compared to 5-fluorouracil (5-FU) and Triamcinolone Acetonide(TAC) for the treatment of Keloids: A Randomized Control Trial | 12 weeks
  The observer scale of the POSAS consists of six items (vascularity, Pigmentation, thickness, relief, pliability and surface area). All items are scored on a scale ranging from
  1 ('like normal skin') to 10 ('worst scar imaginable').The sum of the six items results in a total score of the POSAS observer scale.
efficacy of intralesional bleomycin and combination of triamcinolone acetonide and 5-flourouracil in treating keloids, comparing the scar reduction in accordance with the patient and observer scar (POSAS) scale in two groups. | 4 months
  Efficacy will be assessed by comparing the scar reduction on in accordance with the patient and observer scar (POSAS) scale in two groups. 50% reduction in score from baseline indicates that treatment is affective . It will be assessed at twice weekly interval till 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moravej H, Forghanian A, Dadkhahfar S, Mozafari N. Intralesional bleomycin versus intralesional triamcinolone in the treatment of keloids and hypertrophic scars. Dermatol Ther. 2022 Sep;35(9):e15730. doi: 10.1111/dth.15730. Epub 2022 Aug 3. PMID 35871490
- [Background] Khan HA, Sahibzada MN, Paracha MM. Comparison of the efficacy of intralesional bleomycin versus intralesional triamcinolone acetonide in the treatment of keloids. Dermatol Ther. 2019 Sep;32(5):e13036. doi: 10.1111/dth.13036. Epub 2019 Aug 8. PMID 31361934
- [Background] Bijlard E, Kouwenberg CA, Timman R, Hovius SE, Busschbach JJ, Mureau MA. Burden of Keloid Disease: A Cross-sectional Health-related Quality of Life Assessment. Acta Derm Venereol. 2017 Feb 8;97(2):225-229. doi: 10.2340/00015555-2498. PMID 27378582